CLINICAL TRIAL: NCT04919395
Title: Evaluation of a "Clip" Device Added to the Current Standard Removal of Contraceptive Implant to Improve Stability of the Implant, Shorten Removal Time, and Increase the Ease of Removal
Brief Title: Preliminary Evaluation of a "Clip" Device for Contraceptive Implant Removal
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: On the single day that the study was open, it became clear that modifications to the clip would be required. Only late in 2023 did it become clear that any continuation of the project would require a new trial.
Sponsor: University of Michigan (Other)
Collaborators: VentureWell (Industry)
Responsible Party: Principal Investigator, Carrie Bell, MD, Associate Professor of Obstetrics and Gynecology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00172715
Record Dates: First submitted 2021-05-27; First posted 2021-06-09 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Contraception
Keywords: Nexplanon removal; Medical device
MeSH Terms: interventions — Surgical Instruments

STUDY DESIGN:
Intervention Model Description: Information regarding the planned intervention study model was removed, as the trial did not meet its recruitment goals.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Clip device removal (Experimental)
  Interventions: Device: Clip device for Nexplanon Removal
- Standard of Care removal (Active Comparator)
  Interventions: Procedure: Standard of Care procedure

INTERVENTIONS:
Device: Clip device for Nexplanon Removal — The clip device will be used to assist in the removal procedure to remove the Nexplanon implant from the subject.
  Arms: Clip device removal
Procedure: Standard of Care procedure — The participants Nexplanon will be removed per standard of care.
  Arms: Standard of Care removal

SUMMARY:
This trial is being completed to understand how the study "Clip" device works when assisting clinicians with Nexplanon removals. The study device clips to the skin to hold the implant still and raise the tip of the implant during removal. The study device may improve the process for removing under arm implants by decreasing procedure time and improving the ease and safety of the procedure.

The results from this study will help the researchers understand whether the study device has the potential to simplify the removal procedure and make this form of birth control safer for patients.

ELIGIBILITY:
Inclusion Criteria:

* Currently using Nexplanon and requesting removal
* Qualifies for outpatient removal
* Ability to understand and sign informed consent

Exclusion Criteria:

* Pregnancy
* Any rashes or skin conditions around the insertion site
* Known allergy to lidocaine
* Known allergy to biocompatible plastics or stainless steel

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — This is a study for participants using birth control.
Enrollment: 4 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2021-06-16 (Actual); Study Completion 2021-06-23 (Actual)

PRIMARY OUTCOMES:
Time to remove the contraceptive implant device | During the intervention/procedure/surgery
  The amount of time that it takes to remove the contraceptive implant will be noted for both groups.
Length of incision used for the removal of the single rod contraceptive implant device | During the intervention/procedure/surgery
  This will be recorded for both groups.

SECONDARY OUTCOMES:
Pain based on the Wong-Baker FACES Pain rating scale from the removal of single rod contraceptive | During the intervention/procedure/surgery
  Participants will be asked to rate the pain they experienced during the procedure.
  Subjects will choose the face that best illustrates the pain they experienced during the procedure. Each face corresponds to a value on a 0-10 scale, with a higher score corresponding to more pain.

CONTACTS AND LOCATIONS:
Overall Officials: Carrie Bell, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No